CLINICAL TRIAL: NCT03184337
Title: Women's Lifestyle and Sleep Intervention for Prediabetes and Metabolic Syndrome
Brief Title: Women's Lifestyle Balance Study
Acronym: LB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LB Study
Record Dates: First submitted 2017-05-30; First posted 2017-06-12 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: PreDiabetes; Metabolic Syndrome; Overweight
Keywords: Weight loss; Women; Sleep; Intervention; Diet; Physical activity; Fitbit
MeSH Terms: conditions — Prediabetic State; Metabolic Syndrome; Overweight; Weight Loss; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Control (Active Comparator): Participants in the active control group will receive 8 group sessions of the CDC's PreventT2 program.
  Interventions: Behavioral: CDC's PreventT2 Program
- Experimental (Experimental): Participants in the experimental group will receive 8 group sessions of the CDC's PreventT2 Program with Added Sleep Content designed to extend and improve sleep.
  Interventions: Behavioral: CDC's PreventT2 Program with Added Sleep Content

INTERVENTIONS:
Behavioral: CDC's PreventT2 Program — The PreventT2 program will involve 8 group sessions administered over 3 months. It is a behavioral intervention focused on achieving weight loss by improving nutritional intake and increasing physical activity. It will also include individual biweekly phone calls for 6 months.
  Arms: Active Control
Behavioral: CDC's PreventT2 Program with Added Sleep Content — The CDC's PreventT2 program with added sleep content will involve 8 group sessions administered over 3 months. It is a behavioral intervention focused on achieving weight loss by improving sleep quality and nutritional intake and increasing sleep duration and physical activity. It will also include individual biweekly phone calls for 6 months.
  Arms: Experimental

SUMMARY:
This pilot study aims to determine whether adding a sleep extension and sleep hygiene intervention to an existing lifestyle improvement program improves its efficacy for weight loss in those at risk for diabetes and cardiovascular disease. Half of the participants will receive the Centers for Disease Control's standard PreventT2 program and half of the participants will receive the same program with an additional sleep intervention.

DETAILED DESCRIPTION:
The goal of this pilot study is to determine whether the efficacy of an existing lifestyle improvement program can be increased by adding a sleep extension and sleep hygiene intervention. Improved sleep can improve weight loss through two possible routes: lessening fatigue may potentiate physical activity (PA), and decreasing appetite may potentiate diet improvements. A sample of 24-30 women will be assigned to either the Centers for Disease Control's (CDC's) standard PreventT2 program or the same program with an additional integrated sleep intervention. Both programs will involve 8 group sessions administered over 3 months, and all women will be followed for a total of 6 months. The primary outcome is weight loss, and secondary outcomes include sleep quality and duration, physical activity, caloric intake, and physiological indicators of cardiovascular and diabetes risk (HbA1c, HOMA-IR, lipids, blood pressure). The combined program has the potential to significantly improve weight loss in those at risk for diabetes and cardiovascular disease (CVD).

ELIGIBILITY:
Inclusion Criteria:

* Female (or self-identify as female)
* Age 30-70 years
* BMI 25-38 (or 23-38 if Asian or other Pacific Islander)
* Time in bed <= 7 hours on a typical weeknight
* Meets diagnostic criteria for prediabetes and/or metabolic syndrome

Exclusion Criteria:

* No regular access to telephone or email (for maintaining contact);
* No access to smartphone, tablet, or laptop computer (for using Fitbit);
* Having a condition that limits physical activity, such as brisk walking;
* Having a diagnosis of type 1 or type 2 diabetes or been previously treated with diabetes medications;
* Having a cardiac event or cardiac surgery in the past year;
* Having a metabolic condition that prevents weight loss;
* Working night shift (Midnight - 4 AM)
* Inability to complete the baseline assessment (REDCap survey and Fitbit tracking of activity, diet, and sleep for 7 days)

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only participant's who self-identify as women will be eligible for this pilot study. If it the results are promising, a larger trial with both genders will be pursued.
Enrollment: 26 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change in body mass index | Baseline and 6 weeks, 3 months, and 6 months after start of intervention
  Body mass index is calculated as the participant's body weight divided by the square of their height.

SECONDARY OUTCOMES:
Change in sleep duration (objective) | Baseline and 6 weeks, 3 months, and 6 months after start of intervention
  Nighttime sleep duration will be objectively assessed over 7 days using a Fitbit monitor
Change in sleep quality (self-report) | Baseline and 6 weeks, 3 months, and 6 months after start of intervention
  Pittsburgh Sleep Quality Index (PSQI)
Change in physical activity (objective) | Baseline and 6 weeks, 3 months, and 6 months after start of intervention
  Daily step counts over 7 days using a Fitbit monitor
Change in physical activity (self-report) | Baseline and 6 weeks, 3 months, and 6 months after start of intervention
  International Physical Activity Questionnaire (IPAQ)
Change in caloric intake | Baseline and 6 weeks, 3 months, and 6 months after start of intervention
  Daily calories consumed over 7 days and recorded using a Fitbit monitor
Change in self-reported dietary intake | Baseline and 6 weeks, 3 months, and 6 months after start of intervention
  'Starting the Conversation' will be used to assess self-reported dietary intake
Change in HbA1c | Baseline and 3 months, and 6 months after start of intervention
  HbA1c blood tests will be used to measure average blood glucose levels.
Change in Fasting Plasma Glucose (FPG) | Baseline and 6 weeks, 3 months, and 6 months after start of intervention
  FPG will be used to measure current blood glucose levels
Change in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | Baseline and 6 weeks after start of intervention
  HOMA-IR is calculated from fasting plasma glucose and insulin levels and will be used to measure insulin resistance.
Change in leptin levels | Baseline and 6 weeks after start of intervention
  Leptin levels will be used to measure the hormone that regulates satiety
Change in lipid profile (total cholesterol, LDL, HDL, triglycerides) | Baseline and 6 weeks, 3 months, and 6 months after start of intervention
  A standard lipid panel will be used to measure cardiovascular risk factors
Change in blood pressure | Baseline and 6 weeks, 3 months, and 6 months after start of intervention
  Blood pressure will be used as a measure of cardiovascular risk
Change in waist circumference | Baseline and 6 months after start of intervention
  Waist circumference will be used to measure central adiposity, an indicator of cardiovascular risk.
Change in self-assessed general health | Baseline and 6 weeks, 3 months, and 6 months after start of intervention
  The Promis General Health measure will be used to assess the participant's perception of their general health

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Chesla, RN, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chesla CA, Gay C, Bauer L, Bender MS, Lee K. Preventing Type 2 Diabetes Among Midlife Women: A Feasibility Study Comparing a Combined Sleep and Lifestyle Intervention With a Standard Lifestyle Intervention. Diabetes Educ. 2020 Oct;46(5):424-434. doi: 10.1177/0145721720943128. Epub 2020 Aug 6. PMID 32757824